CLINICAL TRIAL: NCT06381726
Title: Personalized Rendering of Motor System Functional Plasticity Potential to Improve Glioma Resection and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Lorenzo Bello, Full Professor, University of Milan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Progetto AIRC IG-2022 ID 27184
Record Dates: First submitted 2024-03-28; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Glioma; Glioma, Malignant
Keywords: Glioma; Neurosurgery; Chemotherapy, Neoadjuvant; Motor Rehabilitation; Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging; Resting State Functional Magnetic Resonance Imaging; Functional Magnetic Resonance Imaging; Functional Connectomics; Structural Connectomics; Neuronal Plasticity; Higher Nervous Activity; Neurological Rehabilitation; Antineoplastic Protocols
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: Patients immediately candidate for resection will be assessed neurologically, neuropsychologically and by functional MRI. Extent of resection will be assessed on <48hrs and 2-month MRI. Neurological and neuropsychological assessment will be performed during regular follow-up. Patients not requiring an adjuvant treatment according to tumor board meeting will be submitted to functional MRI at 4-8 and 12 months from surgery. Patients not immediately eligible for resection will be submitted to biopsy for histomolecular definition. Patients not requiring radiation therapy will be submitted to neurological, neuropsychological, and functional MRI evaluation. Upon clinical context, patients will undergo motor rehabilitation and/or chemotherapy. After 3-6 months, patients will undergo functional MRI and evaluated for surgery. Neurological and neuropsychological evaluation will be performed at treatment initiation, every month during treatment, at admission for surgery and 1 month after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Spontaneous motor reorganization: observation (Active Comparator): Only neurological and neuropsychological assessment as per normal clinical routine and conventional and advanced functional, resting-state MRI acquisitions
  Interventions: Diagnostic Test: Resting State Functional Magnetic Resonance Imaging (rs-fMRI)
- Enhanced motor reorganization: upfront Motor Rehabilitation (Experimental): Patients submitted to motor rehabilitation program aimed at learning unimanual and bimanual coordinated sequences, along with personalized exercise according to tumor location (frontal vs parietal). For 6 months each patient will perform the motor training program in outpatient training session, checked by a physiotherapist for corrected execution at home 3 times/week, and is assessed for the correct training execution and progresses in training sessions each month, by physical therapists at the Rehabilitation Unit and on a weekly schedule by on-line distant monitoring (telemedicine).
  Interventions: Behavioral: Up-front Motor Rehabilitation
- Enhanced motor reorganization: upfront Chemotherapy (Experimental): Temozolomide-based regimen of 6 months duration is applied. Treatment will be discontinued in case of toxicity (G2-G4).
  Interventions: Drug: Up-front Chemotherapy
- Enhanced motor reorganization: upfront Chemotherapy + Motor Rehabilitation (Experimental): Temozolomide-based regimen of 6 months duration is applied. Treatment will be discontinued in case of toxicity (G2-G4).
  Patients will also be submitted to motor rehabilitation program aimed at learning unimanual and bimanual coordinated sequences, along with personalized exercise according to tumor location (frontal vs parietal). For 6 months each patient will perform the motor training program in outpatient training session, checked by a physiotherapist for corrected execution at home 3 times/week, and is assessed for the correct training execution and progresses in training sessions each month, by physical therapists at the Rehabilitation Unit and on a weekly schedule by on-line distant monitoring (telemedicine).
  Interventions: Behavioral: Up-front Motor Rehabilitation; Drug: Up-front Chemotherapy

INTERVENTIONS:
Diagnostic Test: Resting State Functional Magnetic Resonance Imaging (rs-fMRI) — rs-fMRI + neurological and neuropsychological evaluation at preoperative timepoint and 1-2 months postop, 3-4 months postop, 6-8 months postop, 12 months postop
  Arms: Spontaneous motor reorganization: observation
Behavioral: Up-front Motor Rehabilitation — personalized motor rehabilitation for 6 months + rs-fMRI + neurological and neuropsychological evaluation before starting motor rehabilitation, at 2-3 months during rehabilitation, 6-9 months during rehabilitation, before surgery (if surgery indicated by tumour board), 1 month postop, 2-3 months postop
  Arms: Enhanced motor reorganization: upfront Chemotherapy + Motor Rehabilitation; Enhanced motor reorganization: upfront Motor Rehabilitation
Drug: Up-front Chemotherapy — Temozolomide at either 6 cycles consisting of 150-200 mg per square meter for 5 days during each 28-day cycle, or metronomic schedule, + rs-fMRI + neurological and neuropsychological evaluation before starting motor rehabilitation, at 2-3 months during rehabilitation, 6-9 months during rehabilitation, before surgery (if surgery indicated by tumour board), 1 month postop, 2-3 months Post
  Arms: Enhanced motor reorganization: upfront Chemotherapy; Enhanced motor reorganization: upfront Chemotherapy + Motor Rehabilitation

SUMMARY:
Background Lower-grade-gliomas affect young patients, thus the longest progression-free-survival (PFS) with a high level quality of life is crucial. Surgery most significantly impacts on tumor natural history, postponing recurrence, improving symptoms, decreasing the need of adjuvant therapies, with extent of resection, gross-total and supra-total (GTR and STR), strongly associating with longest PFS. Achievement of GTR or STR depends on the degree of functional reorganization induced by glioma. Consequently, a successful treatment fostering neural circuit reorganization before surgery, would increase the chance of GRT/STR.

Hypothesis The plastic potential of motor system suggests that reorganization of circuits controlling hand movements could be presurgically fostered in LGG patients by enhancing plasticity with up-front motor-rehabilitation and/or by decreasing tumor infiltration with up-front chemotherapy. Advanced neuroimaging allows to infer the neuroplasticity potential. Intraoperative assessment of the motor circuits functionality will validate reliability of preoperative analyses.

Aims The project has 4 aims, investigating: A) the presurgical functional (FC) and structural (SC) connectomics of the hand-motor network to picture the spontaneous reorganization and the influence of clinical, imaging and histomolecular variables; B) the dynamic of FC and SC after tumor resection; C) changes in FC and SC maps after personalized upfront motor rehabilitation and/or chemotherapy; D) the effect of FC and SC upfront treatment on the achievement of GTR/STR preserving hand dexterity.

Experimental Design Resting-state fMRI and diffusion-MRI will provide FC and SC maps pre- and post-surgery; personalized up-front motor rehabilitation and/or chemotherapy will be administered; Intraoperative brain mapping procedures will generate data to validate the maps.

Expected Results

1. Provide a tool to render the motor functional reorganization predictive of surgical outcome.
2. Identify demographic, clinical and imaging variables associated with functional reorganization.
3. Describe the gain induced by up-front treatment.
4. Distinguish "patterns" predicting chance for GTR/STR from "patterns" suggesting need for up-front treatment.

Impact On Cancer Results will increase the achievement of GTR/STR, preserving motor integrity, with dramatic impact on LGGs natural history.

ELIGIBILITY:
Inclusion Criteria (ARM 1):

* Patients signing informed consent for participation in the study
* Males and females
* Age ≥ 18 years
* Patients with lower-grade gliomas with involvement of the motor pathways who are candidates for surgery

Inclusion Criteria (ARM 2/3/4):

* Patients signing informed consent for participation in the study
* Males and females
* Age ≥ 18 years
* Patients with lower-grade gliomas treated over two years with tumors only biopsied and/or partially resected and eligible for second surgery

Exclusion Criteria:

* Age <18 years
* Inability to adhere to standard study controls
* Subjects unable to understand and freely provide consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Muscle power | ARM 1: preop, 1-2 months postop, 3-4 months postop, 6-8 months postop, 12 months postop; ARM 2/3/4: before starting treatment, at 2-3 and 6-9 months during treatment, before surgery (if indicated), 1 month postop, 2-3 months postop
  MRC Muscle power assessment (0-5)
Motor praxia | ARM 1: preop, 1-2 months postop, 3-4 months postop, 6-8 months postop, 12 months postop; ARM 2/3/4: before starting treatment, at 2-3 and 6-9 months during treatment, before surgery (if indicated), 1 month postop, 2-3 months postop
  ARAT test (Grasp, Grip, Pinch, each consisting of 3 items scoring 0 [not performed, 1/2 abnormal, 3 ok]), De Renzi test (24 complex gestures with individual scoring 0-3 [0 no execution/always abnormal, 2/1 ok after 1 or 2 trials, 3 ok] each evaluating one or more among finger movements [total score 0-36], hand movements [total score 0-36], hand and finger position [total score 0-36], sequence of movements [total score 0-36], meaningful gestures [total score 0-36], meaningless gestures [total score 0-36]; tool pantomime for 10 objects individual score 0 if always incorrect, 1 if correct after command repetition, 2 correct immediately, total score range 0-20)

SECONDARY OUTCOMES:
Comprehensive neuropsychological assessment | ARM 1: preop, 1-2 months postop, 3-4 months postop, 6-8 months postop, 12 months postop; ARM 2/3/4: before starting treatment, at 2-3 and 6-9 months during treatment, before surgery (if indicated), 1 month postop, 2-3 months postop
  Language: Naming test; Fhonemic and Semantic Fluency Verbal and Spatial Memory: 15 Rey's Words; Recall Rey figure; Visuo-spatial test: Rey's Copy; Cancellation Test Attention and Executive Functions: Attentive matrice and Trail Making test For each listed test, equivalent score, from 0 to 4, is used.
  Mood Disorders. HADS test (score 0-21 : 0-7= Normal; 8-21 Mood disorders

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Bello, MD, Principal Investigator — University of Milan
Locations (1):
- IRCCS Ospedale Galeazzi Sant'Ambrogio, Milan, Lombardy, Italy

REFERENCES:
- [Background] Bello L, Riva M, Fava E, Ferpozzi V, Castellano A, Raneri F, Pessina F, Bizzi A, Falini A, Cerri G. Tailoring neurophysiological strategies with clinical context enhances resection and safety and expands indications in gliomas involving motor pathways. Neuro Oncol. 2014 Aug;16(8):1110-28. doi: 10.1093/neuonc/not327. Epub 2014 Feb 4. PMID 24500420
- [Background] Castellano A, Donativi M, Ruda R, De Nunzio G, Riva M, Iadanza A, Bertero L, Rucco M, Bello L, Soffietti R, Falini A. Evaluation of low-grade glioma structural changes after chemotherapy using DTI-based histogram analysis and functional diffusion maps. Eur Radiol. 2016 May;26(5):1263-73. doi: 10.1007/s00330-015-3934-6. Epub 2015 Aug 30. PMID 26318368
- [Background] Cochereau J, Deverdun J, Herbet G, Charroud C, Boyer A, Moritz-Gasser S, Le Bars E, Molino F, Bonafe A, Menjot de Champfleur N, Duffau H. Comparison between resting state fMRI networks and responsive cortical stimulations in glioma patients. Hum Brain Mapp. 2016 Nov;37(11):3721-3732. doi: 10.1002/hbm.23270. PMID 27246771
- [Background] Fornia L, Ferpozzi V, Montagna M, Rossi M, Riva M, Pessina F, Martinelli Boneschi F, Borroni P, Lemon RN, Bello L, Cerri G. Functional Characterization of the Left Ventrolateral Premotor Cortex in Humans: A Direct Electrophysiological Approach. Cereb Cortex. 2018 Jan 1;28(1):167-183. doi: 10.1093/cercor/bhw365. PMID 27920095
- [Background] Fornia L, Rossi M, Rabuffetti M, Leonetti A, Puglisi G, Vigano L, Simone L, Howells H, Bellacicca A, Bello L, Cerri G. Direct Electrical Stimulation of Premotor Areas: Different Effects on Hand Muscle Activity during Object Manipulation. Cereb Cortex. 2020 Jan 10;30(1):391-405. doi: 10.1093/cercor/bhz139. PMID 31504261
- [Background] Fornia L, Rossi M, Rabuffetti M, Bellacicca A, Vigano L, Simone L, Howells H, Puglisi G, Leonetti A, Callipo V, Bello L, Cerri G. Motor impairment evoked by direct electrical stimulation of human parietal cortex during object manipulation. Neuroimage. 2022 Mar;248:118839. doi: 10.1016/j.neuroimage.2021.118839. Epub 2021 Dec 25. PMID 34963652
- [Background] Howells H, Puglisi G, Leonetti A, Vigano L, Fornia L, Simone L, Forkel SJ, Rossi M, Riva M, Cerri G, Bello L. The role of left fronto-parietal tracts in hand selection: Evidence from neurosurgery. Cortex. 2020 Jul;128:297-311. doi: 10.1016/j.cortex.2020.03.018. Epub 2020 Apr 10. PMID 32362441
- [Background] Kong NW, Gibb WR, Badhe S, Liu BP, Tate MC. Plasticity of the Primary Motor Cortex in Patients with Primary Brain Tumors. Neural Plast. 2020 Jul 3;2020:3648517. doi: 10.1155/2020/3648517. eCollection 2020. PMID 32714384
- [Background] Puglisi G, Howells H, Sciortino T, Leonetti A, Rossi M, Conti Nibali M, Gabriel Gay L, Fornia L, Bellacicca A, Vigano L, Simone L, Catani M, Cerri G, Bello L. Frontal pathways in cognitive control: direct evidence from intraoperative stimulation and diffusion tractography. Brain. 2019 Aug 1;142(8):2451-2465. doi: 10.1093/brain/awz178. PMID 31347684
- [Background] Raffin E, Siebner HR. Use-Dependent Plasticity in Human Primary Motor Hand Area: Synergistic Interplay Between Training and Immobilization. Cereb Cortex. 2019 Jan 1;29(1):356-371. doi: 10.1093/cercor/bhy226. PMID 30364930
- [Background] Rossi M, Fornia L, Puglisi G, Leonetti A, Zuccon G, Fava E, Milani D, Casarotti A, Riva M, Pessina F, Cerri G, Bello L. Assessment of the praxis circuit in glioma surgery to reduce the incidence of postoperative and long-term apraxia: a new intraoperative test. J Neurosurg. 2019 Jan 1;130(1):17-27. doi: 10.3171/2017.7.JNS17357. Epub 2018 Feb 23. PMID 29473778
- [Background] Rossi M, Ambrogi F, Gay L, Gallucci M, Conti Nibali M, Leonetti A, Puglisi G, Sciortino T, Howells H, Riva M, Pessina F, Navarria P, Franzese C, Simonelli M, Ruda R, Bello L. Is supratotal resection achievable in low-grade gliomas? Feasibility, putative factors, safety, and functional outcome. J Neurosurg. 2019 May 17;132(6):1692-1705. doi: 10.3171/2019.2.JNS183408. Print 2020 Jun 1. PMID 31100730
- [Background] Rossi M, Conti Nibali M, Vigano L, Puglisi G, Howells H, Gay L, Sciortino T, Leonetti A, Riva M, Fornia L, Cerri G, Bello L. Resection of tumors within the primary motor cortex using high-frequency stimulation: oncological and functional efficiency of this versatile approach based on clinical conditions. J Neurosurg. 2019 Aug 9;133(3):642-654. doi: 10.3171/2019.5.JNS19453. Print 2020 Sep 1. PMID 31398706
- [Background] Rossi M, Sciortino T, Conti Nibali M, Gay L, Vigano L, Puglisi G, Leonetti A, Howells H, Fornia L, Cerri G, Riva M, Bello L. Clinical Pearls and Methods for Intraoperative Motor Mapping. Neurosurgery. 2021 Feb 16;88(3):457-467. doi: 10.1093/neuros/nyaa359. PMID 33476393
- [Background] Rossi M, Gay L, Ambrogi F, Conti Nibali M, Sciortino T, Puglisi G, Leonetti A, Mocellini C, Caroli M, Cordera S, Simonelli M, Pessina F, Navarria P, Pace A, Soffietti R, Ruda R, Riva M, Bello L. Association of supratotal resection with progression-free survival, malignant transformation, and overall survival in lower-grade gliomas. Neuro Oncol. 2021 May 5;23(5):812-826. doi: 10.1093/neuonc/noaa225. PMID 33049063
- [Background] Rossi M, Vigano L, Puglisi G, Conti Nibali M, Leonetti A, Gay L, Sciortino T, Fornia L, Callipo V, Lamperti M, Riva M, Cerri G, Bello L. Targeting Primary Motor Cortex (M1) Functional Components in M1 Gliomas Enhances Safe Resection and Reveals M1 Plasticity Potentials. Cancers (Basel). 2021 Jul 28;13(15):3808. doi: 10.3390/cancers13153808. PMID 34359709
- [Background] Sanes JN, Donoghue JP. Plasticity and primary motor cortex. Annu Rev Neurosci. 2000;23:393-415. doi: 10.1146/annurev.neuro.23.1.393. PMID 10845069
- [Background] Simone L, Fornia L, Vigano L, Sambataro F, Rossi M, Leonetti A, Puglisi G, Howells H, Bellacicca A, Bello L, Cerri G. Large scale networks for human hand-object interaction: Functionally distinct roles for two premotor regions identified intraoperatively. Neuroimage. 2020 Jan 1;204:116215. doi: 10.1016/j.neuroimage.2019.116215. Epub 2019 Sep 24. PMID 31557544
- [Background] Southwell DG, Hervey-Jumper SL, Perry DW, Berger MS. Intraoperative mapping during repeat awake craniotomy reveals the functional plasticity of adult cortex. J Neurosurg. 2016 May;124(5):1460-9. doi: 10.3171/2015.5.JNS142833. Epub 2015 Nov 6. PMID 26544767
- [Background] Sun L, Yin D, Zhu Y, Fan M, Zang L, Wu Y, Jia J, Bai Y, Zhu B, Hu Y. Cortical reorganization after motor imagery training in chronic stroke patients with severe motor impairment: a longitudinal fMRI study. Neuroradiology. 2013 Jul;55(7):913-25. doi: 10.1007/s00234-013-1188-z. Epub 2013 Apr 26. PMID 23619700
- [Background] Takeuchi N, Izumi S. Combinations of stroke neurorehabilitation to facilitate motor recovery: perspectives on Hebbian plasticity and homeostatic metaplasticity. Front Hum Neurosci. 2015 Jun 23;9:349. doi: 10.3389/fnhum.2015.00349. eCollection 2015. PMID 26157374
- [Background] van Dokkum LEH, Moritz Gasser S, Deverdun J, Herbet G, Mura T, D'Agata B, Picot MC, Menjot de Champfleur N, Duffau H, Molino F, le Bars E. Resting state network plasticity related to picture naming in low-grade glioma patients before and after resection. Neuroimage Clin. 2019;24:102010. doi: 10.1016/j.nicl.2019.102010. Epub 2019 Oct 24. PMID 31734532
- [Background] Vigano L, Fornia L, Rossi M, Howells H, Leonetti A, Puglisi G, Conti Nibali M, Bellacicca A, Grimaldi M, Bello L, Cerri G. Anatomo-functional characterisation of the human "hand-knob": A direct electrophysiological study. Cortex. 2019 Apr;113:239-254. doi: 10.1016/j.cortex.2018.12.011. Epub 2018 Dec 24. PMID 30708312
- [Background] Vigano L, Howells H, Fornia L, Rossi M, Conti Nibali M, Puglisi G, Leonetti A, Simone L, Bello L, Cerri G. Negative motor responses to direct electrical stimulation: Behavioral assessment hides different effects on muscles. Cortex. 2021 Apr;137:194-204. doi: 10.1016/j.cortex.2021.01.005. Epub 2021 Jan 29. PMID 33640851
- [Background] Vigano L, Howells H, Rossi M, Rabuffetti M, Puglisi G, Leonetti A, Bellacicca A, Conti Nibali M, Gay L, Sciortino T, Cerri G, Bello L, Fornia L. Stimulation of frontal pathways disrupts hand muscle control during object manipulation. Brain. 2022 May 24;145(4):1535-1550. doi: 10.1093/brain/awab379. PMID 34623420
- [Background] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Background] Zhao Z, Wang X, Fan M, Yin D, Sun L, Jia J, Tang C, Zheng X, Jiang Y, Wu J, Gong J. Altered Effective Connectivity of the Primary Motor Cortex in Stroke: A Resting-State fMRI Study with Granger Causality Analysis. PLoS One. 2016 Nov 15;11(11):e0166210. doi: 10.1371/journal.pone.0166210. eCollection 2016. PMID 27846290